CLINICAL TRIAL: NCT02364557
Title: A Phase IIR/III Trial of Standard of Care Therapy With or Without Stereotactic Body Radiotherapy (SBRT) and/or Surgical Ablation for Newly Oligometastatic Breast Cancer
Brief Title: Testing Whether Treating Breast Cancer Metastases With Surgery or High-Dose Radiation Improves Survival
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-BR002; NCI-2014-01810 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BR002; NRG-BR002 (Other: NRG Oncology); NRG-BR002 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2015-02-05; First posted 2015-02-18 (Estimated); Results first posted 2023-02-08 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage IV Breast Cancer American Joint Committee on Cancer (AJCC) v8; Metastatic Breast Carcinoma; Metastatic Malignant Neoplasm in the Bone; Metastatic Malignant Neoplasm in the Liver; Metastatic Malignant Neoplasm in the Lung; Metastatic Malignant Neoplasm in the Lymph Nodes; Metastatic Malignant Neoplasm in the Spine; Prognostic Stage IV Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis | interventions — Radiosurgery; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): Standard of care systemic therapy at the discretion of the treating physician.
- Standard of Care + Ablation (Experimental): Standard of care systemic therapy plus ablation of all metastases by stereotactic body radiotherapy or surgery at the discretion of the treating physician.
  Interventions: Radiation: Stereotactic Body Radiotherapy; Procedure: Surgery

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Patients receive 1, 3, or 5 fractions of radiation, beginning within 6 weeks of study entry.
  * For metastases in the peripheral lung, patients receive a single fraction of 30 Gy or 3 fractions for a total of 45 Gy.
  * For a single liver metastases, patients receive a single fraction of 30 Gy.
  * For metastases in the abdominal-pelvic or liver (>1), patients receive 3 fractions for a total of 45 Gy.
  * For metastases in the central lung or mediastinal/ cervical lymph nodes, patients receive 5 fractions for a total of 50 Gy.
  * For spinal metastases, patients receive 1 fraction of 20 Gy.
  * For non-spinal osseous metastases, patients receive 3 fractions for a total of 30 Gy.
  * For thoracic/cervical spine metastases, patients receive 5 fractions for a total of 35 Gy.
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiosurgery; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery; SBRT; stereotactic ablative radiotherapy (SABR)
  Arms: Standard of Care + Ablation
Procedure: Surgery — All surgical resections will be approached with intent of an R0 resection (rendering the patient with no evidence of measureable disease and pathologic negative margin) and must occur within 6 weeks of study entry. Approach to surgery will be based upon the treating surgeon. An open, laparoscopic, or thorascopic approach is acceptable.
  Arms: Standard of Care + Ablation

SUMMARY:
This randomized phase II/III trial studies how well standard of care therapy with stereotactic radiosurgery and/or surgery works and compares it to standard of care therapy alone in treating patients with breast cancer that has spread to one or two locations in the body (limited metastatic) that are previously untreated. Standard of care therapy comprising chemotherapy, hormonal therapy, biological therapy, and others may help stop the spread of tumor cells. Radiation therapy and/or surgery is usually only given with standard of care therapy to relieve pain; however, in patients with limited metastatic breast cancer, stereotactic radiosurgery, also known as stereotactic body radiation therapy, may be able to send x-rays directly to the tumor and cause less damage to normal tissue and surgery may be able to effectively remove the metastatic tumor cells. It is not yet known whether standard of care therapy is more effective with stereotactic radiosurgery and/or surgery in treating limited metastatic breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Phase II: To determine whether ablation [through stereotactic body radiation therapy (SBRT) (stereotactic radiosurgery) and/or surgical resection of all known metastases] in oligometastatic breast cancer patients provides a sufficient signal for improved progression-free survival (PFS) to warrant full accrual to the Phase III portion of the trial.

II. Phase III: To determine whether ablation (through SBRT and/or surgical resection of all known metastases) in oligometastatic breast cancer patients significantly improves overall survival (OS).

SECONDARY OBJECTIVES:

I. To evaluate treated metastasis control according to tumor receptor status [estrogen receptor (ER), progesterone receptor (PR), human epidermal growth factor receptor 2 (HER2)], use of chemotherapy, surgery versus (vs.) ablative therapy, and number of metastases.

II. To evaluate whether the addition of ablative metastasis directed therapy significantly reduces the number of distant recurrences (new metastases) in patients who progress according to tumor receptor status (ER, PR, HER-2); use of chemotherapy, and number of metastases.

III. To evaluate adverse events in patients who receive ablative metastasis-directed therapy to all known metastases in addition to standard medical therapy compared with those treated with standard medical therapy alone.

EXPLORATORY OBJECTIVE:

I. To explore the most appropriate and clinically relevant technological parameters to ensure quality and effectiveness throughout the radiation therapy processes, including imaging, simulation, target and critical structure definition, treatment planning, image guidance, and delivery.

TRANSLATIONAL RESEARCH OBJECTIVES:

I. To determine whether < 5 circulating tumor cells (CTCs) (per 7.5 ml of blood) is an independent prognostic (outcome) marker for improved PFS and OS in oligometastatic breast cancer.

II. To determine whether < 5 CTCs (per 7.5 ml of blood) is an independent predictive (response to therapy) marker for improved PFS and OS in oligometastatic breast cancer.

III. To determine whether eliminating CTCs (0/7.5 ml of blood in patients with at least 2 CTCs at registration) is both a prognostic and predictive marker for improved PFS and OS.

IV. To evaluate the prognostic and predictive properties of CTC count as a continuous measure of PFS and OS.

V. To store material for retrospective analysis of circulating tumor deoxyribonucleic acid (ctDNA).

VI. To store material for retrospective analysis of circulating micro-ribonucleic acid (RNA).

ELIGIBILITY:
Inclusion Criteria:

* A patient cannot be considered eligible for this study unless all of the following conditions are met.
* Pathologically confirmed metastatic breast cancer
* Known estrogen, progesterone, and HER2 status of either primary tumor or metastasis;

  * Note: estrogen, progesterone and HER2 status of metastasis preferred for stratification
* Number of allowable metastases:

  * =< 4 metastases seen on standard imaging within 60 days prior to registration when all metastatic disease is located within the following sites:

    * Peripheral lung
    * Osseous (bone)
    * Spine
    * Central lung
    * Abdominal-pelvic metastases (lymph node/adrenal gland)
    * Liver
    * Mediastinal/cervical lymph node
* All known disease amenable to metastasis-directed therapy with either SBRT or resection

  * Note: Symptomatic bone metastasis are allowed if ablative therapy can be delivered
  * Note: Sites for possible surgical excision include lung, liver, adrenal gland, bone, small intestine, large intestine, ovary, and amenable nodal disease sites
  * Note: Surgical stabilization is allowed for a metastasis if it is followed by conventionally fractionated external beam radiotherapy
* Maximum diameter of individual metastasis in any dimension =< 5 cm
* There are no restrictions on distance between the metastases
* Patients must be registered within 365 days of the initial metastatic breast cancer diagnosis; first-line standard systemic therapy (chemotherapy, anti-endocrine therapy, anti-HER2, or other standard targeted therapy) for metastatic breast cancer must be given or planned to be given; if given before study entry, it cannot have exceeded a duration of 12 months at the time of registration (Note: sequencing of ablative therapy [surgery or SBRT] relative to systemic therapy, for patients randomized to Arm 2, is at the discretion of the treating physician)
* The primary tumor site must be controlled prior to registration

  * For those who present with synchronous primary and oligometastatic disease, primary must be controlled prior to registration
  * The definition of control is definitive surgery by excision or mastectomy (+/- radiotherapy) per institution preference For those who present with local recurrence and oligometastatic disease, local recurrence must be controlled prior to registration
  * The definition of control is definitive surgery by excision or mastectomy (+/- radiotherapy) per institution preference
* Appropriate stage for study entry based on the following diagnostic workup:

  * History/physical examination within 60 days prior to registration
  * Clinical grade computed tomography (CT) scans of the chest, abdomen, and pelvis with radionuclide bone scan OR whole body positron emission tomography (PET)/CT within 60 days prior to study registration
* Zubrod performance status =< 2 within 60 days prior to registration
* Blood cell count (CBC)/differential obtained within 60 days prior to registration on study
* Absolute neutrophil count (ANC) >= 500 cells/mm^3
* Platelets >= 50,000 cells/mm^3
* Hemoglobin >= 8.0 g/dl (note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
* For females of child-bearing potential, negative serum or urine pregnancy test within 14 days prior to study registration
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Patients with any of the following conditions are NOT eligible for this study.
* Pathologic evidence of active primary disease or local/regional breast tumor recurrence at the time of registration;
* Co-existing or prior invasive malignancy (except non-melanomatous skin cancer), unless disease free for a minimum of 3 years; previous RT dose, date, fraction size, must be reported
* Metastases with indistinct borders making targeting not feasible

  * Note: A potential issue with bone metastases is that they often are not discrete; since many patients on this protocol will have bone metastases, this will be an important issue; theoretically, Houndsfield units might provide an appropriate measure; however, a sclerotic lesion against dense cortical bone will not have a sharp demarcation based on Houndsfield units (HU); therefore, we acknowledge that such determinations will pose a challenge and thus the physician's judgment will be required
* Prior palliative radiation treatment for metastatic disease to be treated on the protocol (including radiopharmaceuticals)
* Metastases located within 3 cm of the previously irradiated structures:

  * Spinal cord previously irradiated to > 40 Gy (delivered in =< 3 Gy/fraction)
  * Brachial plexus previously irradiated to > 50 Gy (delivered in =< 3 Gy/fraction)
  * Small intestine, large intestine, or stomach previously irradiated to > 45 Gy (delivered in =< 3 Gy/fraction)
  * Brainstem previously irradiated to > 50 Gy (delivered in =< 3 Gy/fraction)
  * Whole lung previously irradiated with prior percent volume receiving greater than or equal to 20 Gy (V20Gy)> 30% (delivered in =< 3 Gy/fraction)
  * Primary tumor irradiated with SBRT
  * Metastasis irradiated with SBRT
* Brain metastases
* Exudative, bloody, or cytological proven malignant effusions
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
* Pregnancy; lactating females must cease expression of milk prior to signing consent to be eligible
* Human immunodeficiency virus (HIV) positive with cluster of differentiation (CD)4 count < 200 cells/microliter; note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a cluster of differentiation 4 (CD4) count >= 200 cells/microliter within 30 days prior to registration; note also that HIV testing is not required for eligibility for this protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2014-12-24 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Chmura, Principal Investigator — NRG Oncology
Locations (165):
- United States (154):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Naval Medical Center -San Diego, San Diego, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Saint Joseph's Medical Center, Stockton, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Helen F Graham Cancer Center, Newark, Delaware
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Ascension Saint Vincent Anderson, Anderson, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - GenesisCare USA - Troy, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Virtua Memorial, Mount Holly, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Rex Hematology Oncology Associates-Cary, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Rex Hematology Oncology Associates-Garner, Garner, North Carolina
  - Rex Hematology Oncology Associates-Blue Ridge, Raleigh, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - UNC Rex Cancer Center of Wakefield, Raleigh, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Self Regional Healthcare, Greenwood, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Texas Oncology-Austin Midtown, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Ogden Regional Medical Center, Ogden, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia
- Yonsei University Health System-Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Petrelli F, Ghidini A, Ghidini M, Bukovec R, Trevisan F, Turati L, Indini A, Seghezzi S, Lonati V, Moleri G, Tomasello G, Zaniboni A. Better survival of patients with oligo- compared with polymetastatic cancers: a systematic review and meta-analysis of 173 studies. F1000Res. 2021 May 27;10:423. doi: 10.12688/f1000research.52546.4. eCollection 2021. PMID 35602670

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care + Ablation: Standard of care systemic therapy plus ablation of all metastases by stereotactic body radiotherapy or surgery at the discretion of the treating physician.
  Stereotactic Body Radiotherapy: Patients receive 1, 3, or 5 fractions of radiation, beginning within 6 weeks of study entry.
  * For metastases in the peripheral lung, patients receive a single fraction of 30 Gy or 3 fractions for a total of 45 Gy.
  * For a single liver metastases, patients receive a single fraction of 30 Gy.
  * For metastases in the abdominal-pelvic or liver (>1), patients receive 3 fractions for a total of 45 Gy.
  * For metastases in the central lung or mediastinal/ cervical lymph nodes, patients receive 5 fractions for a total of 50 Gy.
  * For spinal metastases, patients receive 1 fraction of 20 Gy.
  * For non-spinal osseous metastases, patients receive 3 fractions for a total of 30 Gy.
  * For thoracic/cervical spine metastases, patients receive 5 fractions for a total of 35 Gy.
  Surgery: All surgical resections will be approached with intent of an R0 resection (rendering the patient with no evidence of measureable disease and pathologic negative margin) and must occur within 6 weeks of study entry. Approach to surgery will be based upon the treating surgeon. An open, laparoscopic, or thorascopic approach is acceptable.
Period: Overall Study
Arm/Group | Standard of Care (SOC) | Standard of Care + Ablation
Started | 68 | 61
Eligible Population | 65 | 60
AE Population (Eligible and received systemic therapy and/or ablation.) | 62 | 57
Circulating Tumor Cells (CTC) Population (Eligible with blood collection consent and baseline CTC data) | 36 | 26
Completed (Participants contributing data to results are considered to have completed the study.) | 65 | 60
Not Completed | 3 | 1
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) | Standard of Care + Ablation | Total
Number analyzed (Participants) | 65 | 60 | 125
Age, Continuous [Median (Full Range); unit: years] | 53 [32 to 87] | 55.5 [28 to 88] | 54 [28 to 88]
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 years | 24 | 22 | 46
  50-59 years | 19 | 10 | 29
  60-69 years | 15 | 17 | 32
  70-79 years | 5 | 10 | 15
  ≥ 80 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 60 | 125
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 54 | 52 | 106
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 3 | 8
  White | 51 | 45 | 96
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 6 | 3 | 9
Zubrod Performance Status [Count of Participants; unit: Participants] — 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 41 | 41 | 82
    1 | 24 | 19 | 43
Human epidermal growth factor receptor 2 (HER2) status [Count of Participants; unit: Participants] — Positive - breast cancer cells have a lot of HER2 protein. These cancers tend to grow and spread faster than breast cancers that are HER2-negative, but are much more likely to respond to treatment with drugs that target the HER2 protein.
  Negative - breast cancer cells have little or no HER2 protein.
  Participants
    Positive | 8 | 8 | 16
    Negative | 57 | 52 | 109
Estrogen Receptor (ER) Status [Count of Participants; unit: Participants] — Positive - breast cancer cells may need estrogen to grow, these cells may stop growing or die when treated with substances that block the binding and actions of estrogen.
  Negative - breast cancer cells do not need estrogen to grow.
  Participants
    Positive | 58 | 51 | 109
    Negative | 7 | 9 | 16
Progesterone Receptor (PR) Status [Count of Participants; unit: Participants] — Positive - breast cancer cells may need progesterone to grow, these cells may stop growing or die when treated with substances that block the binding and actions of progesterone.
  Negative - breast cancer cells do not need progesterone to grow.
  Participants
    Positive | 35 | 31 | 66
    Negative | 30 | 29 | 59
Hormone Receptor Status [Count of Participants; unit: Participants] — ER- and PR- = breast cancers have no estrogen or progesterone receptors. Treatment with hormone therapy drugs is not helpful for these cancers.
  Participants
    ER+ and/or PR+ | 58 | 54 | 112
    ER- and PR- | 7 | 6 | 13
Patient Metastasis Count [Count of Participants; unit: Participants] — Number of metastases seen on standard imaging prior to enrollment.
  Participants
    1 | 39 | 36 | 75
    >1 | 26 | 24 | 50
First-line standard systemic chemotherapy [Count of Participants; unit: Participants] — Chemotherapy given prior to enrollment.
  Participants
    No | 19 | 16 | 35
    Yes | 46 | 44 | 90
Timing of the diagnosis of the oligometastatic breast disease relative to the primary breast cancer [Count of Participants; unit: Participants] — Synchronous = the diagnosis of oligometastatic breast disease is within 6 months of the primary breast cancer diagnosis.
  Not synchronous = the diagnosis of oligometastatic breast disease is more than 6 months after the primary breast cancer diagnosis.
  Participants
    Synchronous | 12 | 15 | 27
    Not synchronous | 52 | 45 | 97
    Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (Phase II)
Description: Progression (failure) is defined as any of the following: progression of metastases, new metastases, or death. Progression-free survival (PFS) time is defined as time from randomization to the date of first progression, death, or last contact when participant had a documented clinical assessment (censored). PFS rates are estimated using the Kaplan-Meier method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Median PFS is provided.
Time Frame: From randomization to last follow-up. Follow-up schedule: 3 mos after randomization and every 3 months to 24 months, then every six months to five years, then annually. Maximum follow-up at time of analysis was 63 months.
Population: Eligible participants
Measure: Median (70% Confidence Interval); unit: months
Groups:
- Standard of Care + Ablation: Standard of care systemic therapy plus ablation of all metastases by stereotactic body radiotherapy or surgery at the discretion of the treating physician.
  Stereotactic Body Radiotherapy (SBRT): Patients receive 1, 3, or 5 fractions of radiation, beginning within 6 weeks of study entry.
  * For metastases in the peripheral lung, patients receive a single fraction of 30 Gy or 3 fractions for a total of 45 Gy.
  * For a single liver metastases, patients receive a single fraction of 30 Gy.
  * For metastases in the abdominal-pelvic or liver (>1), patients receive 3 fractions for a total of 45 Gy.
  * For metastases in the central lung or mediastinal/ cervical lymph nodes, patients receive 5 fractions for a total of 50 Gy.
  * For spinal metastases, patients receive 1 fraction of 20 Gy.
  * For non-spinal osseous metastases, patients receive 3 fractions for a total of 30 Gy.
  * For thoracic/cervical spine metastases, patients receive 5 fractions for a total of 35 Gy.
  Surgery: All surgical resections will be approached with intent of an R0 resection (rendering the patient with no evidence of measureable disease and pathologic negative margin) and must occur within 6 weeks of study entry. Approach to surgery will be based upon the treating surgeon. An open, laparoscopic, or thorascopic approach is acceptable.
Arm/Group | Standard of Care (SOC) | Standard of Care + Ablation
Number analyzed (Participants) | 65 | 60
months | 23.0 [18.0 to 29.2] | 19.5 [17.0 to 35.6]
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs Standard of Care + Ablation; Assuming an increase in median PFS from 10.5 to 19 months (HR: 0.55), 69 events provide >90% power to conclude superiority with 1-sided α = 0.15; Test type: Superiority; p = 0.36, Log Rank — One-side significance level = 0.15; Hazard Ratio (HR) = 0.92, 70% CI 2-sided [0.71 to 1.17] — Reference level = SOC arm

2. Primary Outcome: Overall Survival (Phase III)
Description: Overall survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored).
Time Frame: From randomization to last follow-up. Follow-up schedule: 3 mos after randomization and every 3 months to 24 months and then annually. Maximum follow-up at time of analysis was 63 months.
Population: It is pre-specified in the study protocol that analysis of Phase III data will not be performed as per the results of the Phase II analysis.
Groups:
- Standard of Care: Standard of care systemic therapy at the discretion of the treating physician.
Arm/Group | Standard of Care | Standard of Care + Ablation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With Treated Metastasis Progression on the SOC + Ablation Arm
Description: Metastasis progression (failure) is defined as the clearance and subsequent recurrence or the development of new metastases in the treated area. Failure time is defined as time from randomization to the date of first failure, last contact when participant had a documented clinical assessment (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method. Two-year failure rates are provided here.
Time Frame: From randomization to last follow-up. Follow-up schedule: 3 months after randomization, every 3 months up to 24 months, every six months up to five years, then annually. Maximum follow-up at time of analysis was 63 months. Two-year rates are provide here.
Population: Eligible participants on the SOC + Ablation arm
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard of Care + Ablation
Number analyzed (Participants) | 60
percentage of participants | 45.0 [29.8 to 59.1]

4. Secondary Outcome: Percentage of Participants With New Metastases
Description: New metastases (failure) is defined as the appearance of any new metastases. Failure time is measured from randomization to the date of first failure, last contact when participant had a documented clinical assessment (censored), or death without failure (competing risk). Failure rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. Two-year failure rates are provided here
Time Frame: From randomization to last follow-up. Follow-up schedule: 3 months after randomization, every 3 months up to 24 months, every six months up to five years, then annually. Maximum follow-up at time of analysis was 63 months.Two-year rates are provided here.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard of Care | Standard of Care + Ablation
Number analyzed (Participants) | 65 | 60
percentage of participants | 47.7 [33.9 to 60.2] | 49.6 [33.9 to 63.5]
Statistical Analysis 1: Comparison: Standard of Care vs Standard of Care + Ablation; Test type: Superiority; p = 0.91, Gray's test — Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.59 to 1.61] — Reference level = SOC arm

5. Secondary Outcome: Number of Patients by Highest Grade Adverse Event Reported
Description: Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From randomization to last follow-up. Follow-up schedule: Arm 1: 3 mos. after randomization / Arm 2: weekly during SBRT and the last day of SBRT; both arms: then every 3 mos. to 24 mos., then annually. Maximum follow-up at time of analysis was 63 months.
Population: Eligible participants who received systemic therapy and/or ablation.
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care (Arm 1): Standard of care systemic therapy at the discretion of the treating physician.
- Standard of Care + Ablation (Arm 2): Standard of care systemic therapy plus ablation of all metastases by stereotactic body radiotherapy or surgery at the discretion of the treating physician.
  Stereotactic Body Radiotherapy: Patients receive 1, 3, or 5 fractions of radiation, beginning within 6 weeks of study entry.
  * For metastases in the peripheral lung, patients receive a single fraction of 30 Gy or 3 fractions for a total of 45 Gy.
  * For a single liver metastases, patients receive a single fraction of 30 Gy.
  * For metastases in the abdominal-pelvic or liver (>1), patients receive 3 fractions for a total of 45 Gy.
  * For metastases in the central lung or mediastinal/ cervical lymph nodes, patients receive 5 fractions for a total of 50 Gy.
  * For spinal metastases, patients receive 1 fraction of 20 Gy.
  * For non-spinal osseous metastases, patients receive 3 fractions for a total of 30 Gy.
  * For thoracic/cervical spine metastases, patients receive 5 fractions for a total of 35 Gy.
  Surgery: All surgical resections will be approached with intent of an R0 resection (rendering the patient with no evidence of measureable disease and pathologic negative margin) and must occur within 6 weeks of study entry. Approach to surgery will be based upon the treating surgeon. An open, laparoscopic, or thorascopic approach is acceptable.
Arm/Group | Standard of Care (Arm 1) | Standard of Care + Ablation (Arm 2)
Number analyzed (Participants) | 62 | 57
Participants
  Grade 1 | 7 | 15
  Grade 2 | 32 | 26
  Grade 3 | 12 | 11
  Grade 4 | 4 | 0

6. Secondary Outcome: Progression-free Survival in the Presence or Absence of Circulating Tumor Cells (CTCs)
Description: The presence of CTCs is defined as ≥ 5 CTCs (per 7.5ml of blood). Progression (failure) is defined as any of the following: progression of metastases, new metastases, or death. Progression-free survival (PFS) time is defined as time from randomization to the date of first progression, death, or last contact when participant had a documented clinical assessment (censored). PFS rates are estimated using the Kaplan-Meier method. The protocol specifies that the distributions of failure times be compared between the groups, which is reported in the statistical analysis results. Two-year PFS rates are provided here
Time Frame: as for outcome 4
Population: Eligible with blood collection consent and baseline CTC data. The protocol specifies that participants from both treatment arms are combined for this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CTCs Absent: < 5 CTCs (per 7.5ml of blood)
- CTCs Present: ≥ 5 CTCs (per 7.5ml of blood)
Arm/Group | CTCs Absent | CTCs Present
Number analyzed (Participants) | 36 | 26
percentage of participants | 42.3 [24.7 to 59.9] | 42.3 [21.8 to 62.9]
Statistical Analysis 1: Comparison: CTCs Absent vs CTCs Present; Test type: Superiority; p = 0.90, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.54 to 2.02] — Reference level = CTCs Absent

ADVERSE EVENTS:
Time Frame: From randomization to last follow-up. Follow-up schedule: Arm 1: 3 months after randomization / Arm 2: weekly during SBRT and the last day of SBRT; then every 3 months to 24 months, then annually. Maximum follow-up at time of analysis was 63 months.
Description: All-cause mortality was assessed in eligible participants. Adverse events were assessed in eligible participants who received systemic therapy and/or ablation.
Arm/Group | Standard of Care (Arm 1) | Standard of Care + Ablation (Arm 2)
All-Cause Mortality (participants affected / at risk) | 18/65 | 17/60
Serious Adverse Events (participants affected / at risk) | 5/62 | 2/57
Other Adverse Events (participants affected / at risk) | 55/62 | 50/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (Arm 1) (N=62) | Standard of Care + Ablation (Arm 2) (N=57)
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1
Hot flashes (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (Arm 1) (N=62) | Standard of Care + Ablation (Arm 2) (N=57)
Anemia (Blood and lymphatic system disorders) | 8 | 8
Blurred vision (Eye disorders) | 4 | 1
Dry eye (Eye disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 7
Constipation (Gastrointestinal disorders) | 8 | 10
Diarrhea (Gastrointestinal disorders) | 14 | 8
Dry mouth (Gastrointestinal disorders) | 4 | 5
Dysphagia (Gastrointestinal disorders) | 4 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 5
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 | 4
Mucositis oral (Gastrointestinal disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 18 | 18
Vomiting (Gastrointestinal disorders) | 6 | 8
Edema limbs (General disorders) | 8 | 3
Fatigue (General disorders) | 40 | 28
General disorders and administration site conditions - Other, specify (General disorders) | 3 | 5
Localized edema (General disorders) | 0 | 4
Non-cardiac chest pain (General disorders) | 4 | 4
Pain (General disorders) | 23 | 9
Infections and infestations - Other, specify (Infections and infestations) | 2 | 6
Skin infection (Infections and infestations) | 5 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 4
Alanine aminotransferase increased (Investigations) | 8 | 6
Alkaline phosphatase increased (Investigations) | 3 | 4
Aspartate aminotransferase increased (Investigations) | 7 | 5
Lymphocyte count decreased (Investigations) | 4 | 7
Neutrophil count decreased (Investigations) | 9 | 9
Platelet count decreased (Investigations) | 7 | 3
Weight gain (Investigations) | 7 | 3
Weight loss (Investigations) | 5 | 0
White blood cell decreased (Investigations) | 11 | 8
Anorexia (Metabolism and nutrition disorders) | 3 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 5
Hypokalemia (Metabolism and nutrition disorders) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 12
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 4
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 8 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 11
Dizziness (Nervous system disorders) | 9 | 3
Headache (Nervous system disorders) | 12 | 6
Peripheral motor neuropathy (Nervous system disorders) | 4 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 19 | 5
Anxiety (Psychiatric disorders) | 12 | 7
Depression (Psychiatric disorders) | 11 | 9
Insomnia (Psychiatric disorders) | 14 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 4
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6 | 6
Hot flashes (Vascular disorders) | 15 | 7
Hypertension (Vascular disorders) | 14 | 10
Hypotension (Vascular disorders) | 1 | 3
Lymphedema (Vascular disorders) | 4 | 7

LIMITATIONS AND CAVEATS:
The trial completed accrual to the phase II portion and was temporarily closed to accrual on September 13, 2019, pending required follow-up for the full phase II analysis, per the protocol-specified statistical analysis plan. The full phase II primary endpoint analysis was done in December 2021 and did not support reopening accrual to address the phase III research question of overall survival.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT02364557/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT02364557/ICF_002.pdf